CLINICAL TRIAL: NCT06856343
Title: REBECCA Real-world Early BrEast CanCer mAnagement REBECCA. a French National Multicentric Real-world Study of Early Breast Cancer Patients
Brief Title: REBECCA Real-world Early BrEast CanCer mAnagement
Acronym: REBECCA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00068
Record Dates: First submitted 2024-12-12; First posted 2025-03-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a French observational, national, multicenter prospective cohort study of patients with HER2-negative eBC treated with olaparib at their physician's discretion.

DETAILED DESCRIPTION:
The purpose to this observational study is to evaluate the rate of completion of adjuvant Olaparib treatment for HER2-negative early breast cancer patients in France.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Patient diagnosed with HER2-negative eBC
* Patient about to be initiated with adjuvant Olaparib at their physician's discretion
* Patient has been informed and does not object to participation in the study.

Exclusion Criteria:

* Patient not consenting to participate.
* Patients included in the Early Access Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from about 60 participating sites to reach the target of 126 subjects, with a maximum of 60% of subtype TN overall.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who receive Olaparib for the full treatment duration | 18 months after inclusion
  The primary outcome is the evaluation of the proportion of patients who receive Olaparib for the full treatment duration, described as 12 months of treatment.

SECONDARY OUTCOMES:
BRCA characteristics: Mutation type | 18 months after inclusion
  Regarding BRCA characteristics: Mutation type: Tumoral (if only tumoral testing performed), somatic, germline.
Type of variants | 18 months after inclusion
  Type of variants: BRCA1 and/or BRCA2, PALB2 mutation, presence of other HRR gene mutations, presence of other mutations
Medical history | 18 months after inclusion
  Family and personal history of cancer/type
Time to Olaparib treatment discontinuation | 18 months after inclusion
  Time to Olaparib Treatment Discontinuation (TTD) or death

CONTACTS AND LOCATIONS:
Locations (42):
- France (42):
  - Research Site, Agen
  - Research Site, Argenteuil
  - Research Site, Avignon
  - Research Site, Beauvais
  - Research Site, Beuvry
  - Research Site, Bezannes
  - Research Site, Caen
  - Research Site, Chambray-lès-Tours
  - Research Site, Champigny-sur-Marne
  - Research Site, Clermont-Ferrand
  - Research Site, Compiègne
  - Research Site, Creil
  - Research Site, Dechy
  - Research Site, FORT de France Cedex
  - Research Site, Fréjus
  - Research Site, Gleizé
  - Research Site, Grenoble
  - Research Site, Le Blanc-Mesnil
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Metz-Tessy
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nice
  - Research Site, Osny
  - Research Site, Paris
  - Research Site, Périgueux
  - Research Site, Plérin
  - Research Site, Poitiers
  - Research Site, Rouen
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Doulchard
  - Research Site, Saint-Etienne
  - Research Site, Saint-Grégoire
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Salouël
  - Research Site, Thonon-les-Bains
  - Research Site, Valence